CLINICAL TRIAL: NCT06296017
Title: Effectiveness of Conservative Interventions in the Treatment of Trigger Finger
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Feray Karademir, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEŞH- EK1- 2023-115
Record Dates: First submitted 2024-02-14; First posted 2024-03-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Trigger Finger; Stenosing Tenosynovitis
MeSH Terms: conditions — Trigger Finger Disorder; Tendon Entrapment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Extracorporeal Shock Wave Therapy (Experimental): Extracorporeal Shock Wave Therapy (ESWT for short) application will be performed on A1 pulley at 15 Hz, 1000 shock wave impulses, and 2.0 bar level, for a total of 5 sessions, one week apart.
  Interventions: Other: Experimental: Extracorporeal Shock Wave Therapy
- Trigger Finger Splint (Experimental): A trigger finger splint that immobilizes the MCF joint will be recommended for the splint treatment group. The patient will be asked to use this splint throughout the day for 8 weeks.
  Interventions: Other: Trigger Finger Splint
- Extracorporeal Shock Wave Therapy+Trigger Finger Splint (Experimental): Splint treatment will be applied together with ESWT. ESWT application will be performed on A1 pulley at 15 Hz, 1000 shock wave impulses, and 2.0 bar level, in a total of 5 sessions, one week apart. A trigger finger splint that immobilizes the MCF joint will be recommended for the splint treatment group. The patient will be asked to use this splint throughout the day for 8 weeks.
  Interventions: Other: Extracorporeal Shock Wave Therapy+ Trigger Finger Splint

INTERVENTIONS:
Other: Experimental: Extracorporeal Shock Wave Therapy — Extracorporeal Shock Wave Therapy (ESWT for short) application will be performed on A1 pulley at 15 Hz, 1000 shock wave impulses, and 2.0 bar level, for a total of 5 sessions, one week apart.
  Arms: Extracorporeal Shock Wave Therapy
Other: Trigger Finger Splint — A trigger finger splint that immobilizes the MCF joint will be recommended for the splint treatment group. The patient will be asked to use this splint throughout the day for 8 weeks.
  Arms: Trigger Finger Splint
Other: Extracorporeal Shock Wave Therapy+ Trigger Finger Splint — Extracorporeal Shock Wave Therapy (ESWT for short) application will be performed on A1 pulley at 15 Hz, 1000 shock wave impulses, and 2.0 bar level, for a total of 5 sessions, one week apart. Also, A trigger finger splint that immobilizes the MCF joint will be recommended.
  Arms: Extracorporeal Shock Wave Therapy+Trigger Finger Splint

SUMMARY:
There is no study in the literature comparing the effectiveness of ESWT and splint therapy, which are the most commonly used approaches in the treatment of Trigger Finger (TF). The aim in this study is to investigate the effectiveness of ESWT and splint therapy used in the treatment of TF.

DETAILED DESCRIPTION:
Volunteer patients who were clinically diagnosed with trigger finger by consulting a doctor at Etlik City Hospital, Hand Surgery Clinic will be included in the randomized controlled prospective study. Patients will be randomly divided into three groups using the 'Random Sequence Generator tab' on Random.org, a randomization website, and different treatment programs will be applied. ESWT application to a group; splint treatment with ESWT to the second group; The third group will receive only splint treatment. ESWT application will be performed on A1 puley at 15 Hz, 1000 shock wave impuls and 2.0 bar level, for a total of 5 sessions, one week apart. In addition to ESWT with the same parameters, a trigger finger splint that immobilizes the MCP joint will be recommended to the ESWT and splint treatment group. The patient will be asked to use this splint throughout the day for 8 weeks. The Splint Group will be offered the same trigger finger splint and will be asked to use it throughout the day for 8 weeks. Evaluation and measurements will be repeated for all three groups before treatment, immediately after treatment (8th week) and 4 weeks after the end of treatment (12th week). The number of individuals to participate in the study was calculated as 54 in total, with 18 people in each group (ESWT Group, ESWT+ Splint Group and Splint Group), according to the power and sample size analysis based on 80% power and 5% Type 1 error rate. Power analysis was performed based on pain intensity as the clinical endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering
* Being between the ages of 18-65
* Being diagnosed with stage 1 or stage 2 (according to the Froimson classification) trigger finger
* Having the language and cognitive skills to answer the questionnaires used in the evaluation

Exclusion Criteria:

* Being pregnant
* Having an inflammatory disorder
* Having had surgery on the hand/wrist
* Having a neurological disease
* NSAIDs, painkillers, etc. being on medication
* De Quervain's tenosynovitis, carpal tunnel syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | pre-treatment and post-treatment at 8 week
  The severity of pain felt by individuals at rest and during challenging activities will be evaluated using the Visual Analog Scale (VAS). The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

SECONDARY OUTCOMES:
Grip and pinch strength | pre-treatment and post-treatment at 8 weeks
  Grip Strength Measurement: Standard, tip, lateral and tripod grip strengths will be performed in the test position standardized by the American Association of Hand Therapists. Jamar hand dynamometer and pinchmeter (Pro Med Products, Atlanta, GA, USA) will be used for evaluation. Grip strength will be measured at the 2nd position of the dynamometer. The evaluation will be made three times for each measurement and the average will be recorded in kg.
Number of trigger | pre-treatment and post-treatment at 8 weeks
  Patients will be asked to open and close their hand ten times and the number of triggers will be recorded out of 10. If the patient's finger becomes locked at any time while making a full fist, they will be asked to stop and a score of 10/10 will be given.
Functional assessment | pre-treatment and post-treatment at 8 weeks
  The Disabilities of the Arm, Shoulder and Hand Questionnaire: DASH contains thirty items regarding symptoms and activities of daily living. The total score is 100, with higher scores indicating more apology.
Treatment satisfaction | pre-treatment and post-treatment at 8 weeks
  Roles and Maudsley Score is used to score treatment satisfaction level. The patient is asked to compare his/her pain level before and after treatment and to indicate whether he or she has benefited.
  1. Excellent: I have no pain, I can do my movements and activities fully, I benefited from the treatment.
  2. Good: I have some discomfort, but I can do my movements and activities fully, my complaints have decreased after the treatment.
  3. Acceptable: My pain level has decreased compared to before the treatment, but I feel discomfort after long-term activities. I received little benefit from the treatment.
  4. Bad: I cannot do activities due to my pain, I did not benefit from the treatment.
Functional assessment | pre-treatment and post-treatment at 8 weeks
  Michigan Hand Outcomes Questionnaire: It consists of six subheadings: general hand function, ADL (unilateral and bilateral), work, pain, aesthetics and satisfaction. Subheadings are filled separately for right and left hands. The score for each title is calculated separately. It is normalized by calculating the percentage of raw scores obtained by summing the scores (0 to 100) given to each question. Higher scores indicate better functional level.

CONTACTS AND LOCATIONS:
Overall Officials: Kadir ÇEVİK, Study Director — Etlik Şehir Hastanesi
Locations (1):
- Feray Karademir, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonnici AV, Spencer JD. A survey of 'trigger finger' in adults. J Hand Surg Br. 1988 May;13(2):202-3. doi: 10.1016/0266-7681_88_90139-8. PMID 3385301
- [Background] Sampson SP, Badalamente MA, Hurst LC, Seidman J. Pathobiology of the human A1 pulley in trigger finger. J Hand Surg Am. 1991 Jul;16(4):714-21. doi: 10.1016/0363-5023(91)90200-u. PMID 1880372
- [Background] Makkouk AH, Oetgen ME, Swigart CR, Dodds SD. Trigger finger: etiology, evaluation, and treatment. Curr Rev Musculoskelet Med. 2008 Jun;1(2):92-6. doi: 10.1007/s12178-007-9012-1. PMID 19468879
- [Background] Flatt AE. Notta's nodules and trigger digits. Proc (Bayl Univ Med Cent). 2007 Apr;20(2):143-5. doi: 10.1080/08998280.2007.11928272. No abstract available. PMID 17431449
- [Background] Froimson A. Tenosynovitis and tennis elbow. Operative hand surgery. 1993:1989-2006.
- [Background] Alsancak S, Güner S, Bilgin S. Efficacy of splinting variations in two different treatment protocols in trigger thumb. JPO: Journal of Prosthetics and Orthotics. 2015;27(1):17-22.
- [Background] Yildirim P, Gultekin A, Yildirim A, Karahan AY, Tok F. Extracorporeal shock wave therapy versus corticosteroid injection in the treatment of trigger finger: a randomized controlled study. J Hand Surg Eur Vol. 2016 Nov;41(9):977-983. doi: 10.1177/1753193415622733. Epub 2016 Sep 28. PMID 26763271